CLINICAL TRIAL: NCT04199689
Title: A Phase 3, International, Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial to Study the Efficacy, Immunogenicity, and Safety of the 9vHPV Vaccine, a Multivalent L1 Virus-like Particle Vaccine, in the Prevention of Oral Persistent Infection With HPV Types 16, 18, 31, 33, 45, 52, or 58 in Adult Males, 20 to 45 Years of Age
Brief Title: Efficacy Against Oral Persistent Infection, Immunogenicity and Safety of the 9-valent Human Papillomavirus Vaccine (9vHPV) in Men Aged 20-45 Years (V503-049)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V503-049; V503-049 (Other: MSD); 205346 (Registry Identifier: JAPIC-CTI); 2022-501974-21 (Registry Identifier: EU CT); U1111-1275-8682 (Registry Identifier: UTN); 2019-003236-23 (EudraCT Number)
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 9vHPV vaccine (Experimental): Single 0.5-mL intramuscular injection at Day 1, Month 2, and Month 6
  Interventions: Biological: 9vHPV Vaccine
- Placebo (Placebo Comparator): Single 0.5-mL intramuscular injection at Day 1, Month 2, and Month 6
  Interventions: Other: Placebo (Saline for Injection)

INTERVENTIONS:
Biological: 9vHPV Vaccine — 9vHPV is an aluminum-adjuvanted recombinant protein vaccine prepared from the highly purified virus-like particles of the recombinant major capsid (L1) protein of HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 given as a 0.5 mL intramuscular injection.
  Other Names: GARDASIL®9; V503
  Arms: 9vHPV vaccine
Other: Placebo (Saline for Injection) — 0.9% sodium chloride given as a 0.5-mL intramuscular injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, immunogenicity and safety of the 9vHPV vaccine in men 20 to 45 years of age. The primary hypothesis tested after the primary database lock is that administration of a 3-dose regimen of 9vHPV vaccine will reduce the incidence of human papillomavirus (HPV) 16/18/31/33/45/52/58-related oral persistent infection (6 months or longer) compared with placebo.

There will also be an Extension Study to offer an opportunity to complete the 3 dose regimen of 9vHPV vaccine for participants who received placebo in the Base Study, or received less than 3 doses of 9vHPV vaccine in the Base Study.

ELIGIBILITY:
Inclusion Criteria:

Base Study:

* Is healthy and is judged to be in good physical health based on medical history and physical examination
* Has provided written informed consent for the study. The participant may also provide consent for future biomedical research. However, the participant may participate in the main study without participating in future biomedical research
* Agrees to provide study personnel with a primary telephone number as well as an alternate means of contact, if available (such as an alternate telephone number or email) for follow-up purposes
* Can read, understand, and complete the electronic vaccination report card (eVRC)
* Has had at least 1 lifetime sexual partner

Extension Study:

* Participants may continue in the Extension Study if Inclusion Criteria #1 and #4 are still met, and the participants was in either the placebo group in the Base Study or the vaccine group in the Base Study but did not complete the vaccination series
* Provides documented consent for the Extension Study

Exclusion Criteria:

Base Study:

* Has a history of HPV-related anal lesion (anal intraepithelial neoplasia or anal cancer) or HPV related head and neck cancer
* Has a history of or clinical evidence at the Day 1 external genital examination of HPV-related external lesion
* Has clinical evidence at the Day 1 external genital examination of gross genital lesion suggesting sexually transmitted disease
* Has a fever (defined as oral temperature ≥100.0°F or ≥37.8°C) within a 24-hour period prior to Day 1 visit
* Has a history of severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention
* Is allergic to any vaccine component, including aluminum, yeast, or BENZONASE®
* Has known thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections
* Is currently immunocompromised or has been diagnosed as having congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition
* Has a history of splenectomy
* Has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate by judgment of investigator
* Is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence at the discretion of the investigator. Alcohol abusers are defined as those who drink despite recurrent social, interpersonal, and/or legal problems because of alcohol use
* Has received within 12 months prior to enrollment, is receiving, or plans to receive during the study, the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide (ARAVA®), TNF-α antagonists, monoclonal antibody therapies (including rituximab [RITUXAN®]), intravenous immunoglobulin (IVIG), anti-lymphocyte sera, or other therapy known to interfere with the immune response. Regarding systemic corticosteroids, a participant will be excluded if he is currently receiving steroid therapy, has recently received such therapy, or has received 2 or more courses of high-dose corticosteroids (≥20 mg/day of prednisone [or equivalent] orally or parenterally) lasting at least 1 week in duration in the year prior. Participants using inhaled, nasal, or topical steroids are considered eligible for the study
* Has received within the 3 months prior to vaccination, is receiving, or plans to receive during the study, any immune globulin product (including RhoGAM™) or blood-derived product other than IVIG
* Has received inactivated or recombinant vaccines within 14 days prior to vaccination or receipt of live vaccines within 21 days prior to vaccination
* Is concurrently enrolled in other clinical studies of investigational agents
* Has previously received a marketed HPV vaccine, or has participated in a clinical trial for any HPV vaccine (receiving either active agent or placebo)
* Has engaged in sexual activity 48 hours prior to vaccination. Sexual activity is defined as: penile penetrative vaginal intercourse with female partner; penile penetrative or receptive anal intercourse with male or female partner; or oral sex involving any contact between participant's mouth with a female partner's vagina, genital or anal area or male partner's penis or genital or anal area. This also includes any contact between participant's partner's mouth with participant's penis, genital or anal area
* Is unlikely to adhere to the study procedures, keep appointments, or is planning to permanently relocate from the area prior to the completion of the study or to leave for an extended period when study visits would need to be scheduled
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study

Extension Study:

- Participants must be excluded from the Extension Study if Base Study Exclusion Criteria #4, 5, 6, 7, 10, 16, or 18 are met

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male participants between the ages of 20 and 45 years (inclusive)
Enrollment: 6033 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2027-08-27 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of HPV 16/18/31/33/45/52/58-related 6-month Persistent Oral Infection | Up to Month 90
  A 6-month persistent infection is defined to have occurred if a participant, after completion of the Month 7 visit, is positive for the same HPV type by the HPV polymerase chain reaction (PCR) assay to at least 1 common gene in Oral Rinse and Gargle (ORG) samples obtained at 2 or more consecutive visits at 6 months (+/-1 month visit window) apart.

SECONDARY OUTCOMES:
Incidence of HPV 6/11-related 6-month Persistent Oral Infection | Up to Month 90
  A 6-month persistent infection is defined to have occurred if a participant, after completion of the Month 7 visit, is positive for the same HPV type by the HPV PCR assay to at least 1 common gene in ORG samples obtained at 2 or more consecutive visits at 6 months (+/-1 month visit window) apart.
Geometric Mean Titers to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 Antibodies | 1 month postdose 3 (Month 7)
  Serum antibodies to HPV types are measured with competitive Luminex immunoassay (cLIA). Geometric mean titers of antibodies to HPV types will be calculated by exponentiating the mean estimates of natural logarithm of the anti-HPV titers.
Percentage of Participants who Seroconvert to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 1 month postdose 3 (Month 7)
  Seroconversion is defined as changing a participant's serostatus from seronegative at Day 1 to seropositive by 4 weeks postdose 3. A participant with anti-HPV cLIA titer at or above the serostatus cutoff of the cLIA for a given HPV type is considered seropositive for that HPV type.
Percentage of Participants with at Least 1 Solicited Injection-site Adverse Event (AE) | Up to 5 days after any vaccination
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. Solicited injection-site AEs such as redness/erythema, swelling, and tenderness/pain at the injection site will be recorded.
Percentage of Participants with Elevated Temperature (Fever) | Up to 5 days after any vaccination
  Participants are asked to record oral body temperatures. The percentage of participants with elevated temperature (≥37.8°C or 100.0°F) will be assessed.
Percentage of Participants Who Report at Least 1 Systemic AE | Up to 15 days after any vaccination
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. Systemic AEs are those not categorized as injection-site AEs.
Percentage of Participants Who Experience at Least 1 Serious Adverse Event (SAE) | Up to 15 days after any vaccination
  A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect, or is another important medical event deemed such by medical or scientific judgment.
Percentage of Participants who Experience at Least 1 Serious Vaccine-Related AE | Up to Month 90
  A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect, or is another important medical event deemed such by medical or scientific judgment. An SAE that is considered by an investigator (a qualified physician) to be vaccine-related will be reported during entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (103):
- United States (32):
  - Valley Clinical Trials Inc. ( Site 0002), Northridge, California
  - Inland Empire Clinical Trials, LLC ( Site 0025), Rialto, California
  - Alta California Medical Group ( Site 0031), Simi Valley, California
  - Encompass Clinical Research ( Site 0028), Spring Valley, California
  - Diablo Clinical Research, Inc ( Site 0042), Walnut Creek, California
  - Clinical Research of South Florida ( Site 0036), Coral Gables, Florida
  - Acevedo Clinical Research Associates ( Site 0001), Miami, Florida
  - Moffitt Cancer Center ( Site 0017), Tampa, Florida
  - Augusta University ( Site 0010), Augusta, Georgia
  - Solaris Clinical Research, LLC ( Site 0003), Meridian, Idaho
  - Cotton-O'Neil Clinical Research Center ( Site 0044), Topeka, Kansas
  - Heartland Research Associates, LLC ( Site 0034), Wichita, Kansas
  - Kentucky Pediatric/Adult Research Inc ( Site 0011), Bardstown, Kentucky
  - Healthcare Research Network LLC ( Site 0035), Hazelwood, Missouri
  - Alliance for Multispecialty Reseach, LLC ( Site 0021), Las Vegas, Nevada
  - Certified Research Associates ( Site 0041), Cortland, New York
  - Laser Surgery Care ( Site 0018), New York, New York
  - Weill Cornell Medicine ( Site 0046), New York, New York
  - Rochester Clinical Research, Inc. ( Site 0008), Rochester, New York
  - PMG Research of Salisbury ( Site 0009), Salisbury, North Carolina
  - Rapid Medical Research, Inc. ( Site 0037), Cleveland, Ohio
  - Preferred Primary Care Physicians ( Site 0032), Pittsburgh, Pennsylvania
  - Coastal Carolina Research Center ( Site 0043), North Charleston, South Carolina
  - Holston Medical Group ( Site 0030), Kingsport, Tennessee
  - University of Texas Medical Branch at Galveston ( Site 0038), Galveston, Texas
  - Texas Center For Drug Development ( Site 0013), Houston, Texas
  - Crossroads Clinical Research LLC ( Site 0027), Victoria, Texas
  - J Lewis Research Inc/Foothill Family Clinic South ( Site 0006), Salt Lake City, Utah
  - J Lewis Research Inc/Jordan River Family Medicine ( Site 0023), South Jordan, Utah
  - Charlottesville Medical Research Center, LLC ( Site 0007), Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0015), Newport News, Virginia
  - Clinical Research Partners, LLC. ( Site 0004), Richmond, Virginia
- Belgium (3):
  - University of Antwerp ( Site 0352), Wilrijk, Antwerpen
  - Universitair Ziekenhuis Gasthuisberg ( Site 0353), Leuven, Vlaams-Brabant
  - Femicare VZW ( Site 0350), Tienen, Vlaams-Brabant
- Brazil (3):
  - Hospital Santo Antonio - Obras Sociais Irma Dulce ( Site 0101), Salvador, Estado de Bahia
  - CPCLIN ( Site 0100), Natal, Rio Grande do Norte
  - Centro de Pesquisa Clinica II - ICHC - FMUSP ( Site 0102), São Paulo
- Colombia (3):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0153), Medellín, Antioquia
  - Clinica de la Costa Ltda. ( Site 0152), Barranquilla, Atlántico
  - Centro de Atención e Investigación Médica SAS - CAIMED CHIA ( Site 0156), Chía, Cundinamarca
- Czechia (4):
  - Centrum ambulantni gynekologie a primarni pece ( Site 0401), Brno, Brno-mesto
  - G-CENTRUM Olomouc s.r.o. ( Site 0400), Olomouc
  - MediStar s.r.o. ( Site 0403), Prague
  - FN Motol ( Site 0402), Prague
- France (5):
  - CHU Dijon Bourgogne - Hopital F. Mitterrand ( Site 0223), Dijon, Cote-d Or
  - Hopital Saint Eloi ( Site 0504), Montpellier, Herault
  - C.H.R.U. de Rennes. Hopital de Pontchaillou ( Site 0507), Rennes, Ille-et-Vilaine
  - CHU Nantes - Hopital Hotel Dieu ( Site 0510), Nantes, Loire-Atlantique
  - Hopital Cochin ( Site 0506), Paris, Île-de-France Region
- Germany (4):
  - Infektiologikum Frankfurt-Sachsenhausen ( Site 0456), Frankfurt am Main, Hesse
  - Epimed GmbH ( Site 0450), Berlin
  - Klinische Forschung Berlin ( Site 0454), Berlin
  - Universitatsklinikum Hamburg-Eppendorf ( Site 0451), Hamburg
- Israel (4):
  - Meir Medical Center ( Site 0602), Kfar Saba, Central District
  - Maccabi Health Services Medical Center ( Site 0604), Tel Aviv, Central District
  - Rambam Medical Center ( Site 0601), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 0600), Jerusalem
- Italy (5):
  - Istittuto Nazionale dei Tumori Regina Elena IRCCS - IFO ( Site 0551), Rome, Roma
  - Azienda Ospedaliera - Universita di Padova ( Site 0555), Padua, Veneto
  - Azienda Ospedaliera Policlinico di Bari ( Site 0550), Bari
  - AOU Policlinico Vittorio Emanuele ( Site 0552), Catania
  - Universita di Roma "La Sapienza" ( Site 0553), Roma
- Japan (15):
  - P-One Clinic, Keikokai Medical Corp. ( Site 1101), Hachiōji, Tokyo
  - Sagiyama Urology Clinic ( Site 1116), Fukuoka
  - Souseikai PS Clinic ( Site 1103), Fukuoka
  - Souseikai Nishikumamoto Hospital ( Site 1104), Kumamoto
  - Medical Corporation Heishinkai OPHAC Hospital ( Site 1105), Osaka
  - Nomura Clinic Namba ( Site 1114), Osaka
  - Medical Corporation Seiwakai Hayakawa Clinic ( Site 1113), Osaka
  - Doujin Memorial Medical Foundation, Meiwa Hospital ( Site 1111), Tokyo
  - Taisei Clinic ( Site 1109), Tokyo
  - Medical Corporation Mori to Umi Tokyo Tokyo Kamata Hospital ( Site 1112), Tokyo
  - Naoko Dermatology Clinic ( Site 1107), Tokyo
  - Medical Corporation Shinanokai Shinanozaka Clinic ( Site 1106), Tokyo
  - Medical Corporation Iseikai My City Clinic ( Site 1108), Tokyo
  - Medical Corporation Houeikai Sekino Clinical Pharmacology Clinic ( Site 1102), Tokyo
  - Kusunoki Clinic ( Site 1110), Tokyo
- Mexico (4):
  - Arke Estudios Clinicos S.A. de C.V. ( Site 0203), Mexico City, Mexico City
  - Instituto Nacional de Salud Publica ( Site 0202), Cuernavaca, Morelos
  - Icaro Investigaciones en Medicina S.A. de C.V. ( Site 0200), Chihuahua City
  - ARKE Estudios Clinicos S.A de C.V ( Site 0211), Veracruz
- Peru (5):
  - Asociacion Civil Selva Amazonica ( Site 0252), Iquitos, Loreto
  - Policlinico Universidad Nacional Mayor de San Marcos ( Site 0257), Lima
  - Investigaciones Medicas en Salud - INMENSA ( Site 0255), Lima
  - Instituto de Investigacion Nutricional - Anexo Huascar ( Site 0251), Lima
  - Asociacion Via Libre ( Site 0250), Lima
- South Korea (5):
  - Korea University Ansan Hospital ( Site 0952), Ansan-si, Kyonggi-do
  - The Catholic University of Korea Eunpyeong St Mary s Hospital ( Site 0954), Seoul
  - Severance Hospital ( Site 0953), Seoul
  - Hallym University Kangnam Sacred Heart Hospital ( Site 0951), Seoul
  - Korea University Guro Hospital ( Site 0950), Seoul
- Spain (3):
  - Institut Catala d Oncologia Hospital Germans Trias i Pujol ( Site 0755), Badalona, Barcelona
  - CAP Centelles ( Site 0751), Centelles, Barcelona
  - ICO L Hospitalet ( Site 0754), L'Hospitalet de Llobregat, Barcelona
- Taiwan (4):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 1003), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 1002), Tainan
  - National Taiwan University Hospital ( Site 1000), Taipei
  - Chang Gung Medical Foundation.Linkou Branch ( Site 1001), Taoyuan District
- Thailand (4):
  - Armed Forces Research Institute of Medical Sciences ( Site 1051), Bangkok, Bangkok
  - Vaccine Trial Center Faculty of Tropical Medicine ( Site 1052), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 1050), Bangkok, Bangkok
  - Research Institute for Health Sciences ( Site 1053), Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Giuliano AR. Initiation of three complementary international studies investigating prevalence of oral HPV infection, burden of HPV-related head and neck disease, and efficacy of 9-valent HPV vaccination against oral HPV persistent infection. Contemp Clin Trials. 2022 Apr;115:106629. doi: 10.1016/j.cct.2021.106629. Epub 2021 Nov 24. No abstract available. PMID 34838718
- [Derived] Morais E, Kothari S, Roberts C, Yen G, Chen YT, Lynam M, Pedros M, Mirghani H, Alemany L, Pavon MA, Waterboer T, Mehanna H, Giuliano AR. Oral human papillomavirus (HPV) and associated factors among healthy populations: The design of the PROGRESS (PRevalence of Oral hpv infection, a Global aSSessment) study. Contemp Clin Trials. 2022 Apr;115:106630. doi: 10.1016/j.cct.2021.106630. Epub 2021 Nov 25. PMID 34838717
- [Derived] Giuliano AR, Wilkin T, Bautista OM, Cheon K, Connor L, Dubey S; Thomas Group; Luxembourg A, Rawat S, Shaw A, Velicer C, Vendetti N, Tu Y. Design of a phase III efficacy, immunogenicity, and safety study of 9-valent human papillomavirus vaccine in prevention of oral persistent infection in men. Contemp Clin Trials. 2022 Apr;115:106592. doi: 10.1016/j.cct.2021.106592. Epub 2021 Oct 19. PMID 34678491
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26203&tenant=MT_MSD_9011